CLINICAL TRIAL: NCT04126408
Title: Safety and Efficacy of Non-invasive Vagus Nerve Stimulation in the Treatment of Headache in Subarachnoid Hemorrhage
Acronym: VANQUISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Tania Rebeiz, Assistant Professor, MD, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-0837
Record Dates: First submitted 2019-09-13; First posted 2019-10-15 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham arm (Sham Comparator): gammaCore sham device which will not provide stimulation of the vagus nerve
  Interventions: Device: gammaCore
- Treatment group (Active Comparator): Active gammaCore device that supplies non-invasive stimulation of the cervical branch of the Vagus nerve
  Interventions: Device: gammaCore

INTERVENTIONS:
Device: gammaCore — The intervention consists of a transcutaneous non-invasive stimulation of the cervical branch of the vagus nerve (nVNS) using gammaCore, an FDA approved device for the treatment of migraine and cluster headache. This will be compared to the sham device, which is the same device which will not provide stimulation to the nerve. Stimulation frequency will be identical to the frequency used in previous nVNS studies for the treatment of migraine headache.

SUMMARY:
This is a single site, randomized, sham-controlled, double blinded pilot study assessing the feasibility, safety, tolerability, and efficacy of non-invasive VNS (nVNS), gammaCore, in the treatment of headache in subarachnoid hemorrhage (SAH). 40 participants will be enrolled, 20 in the active device arm and 20 in the sham arm. The primary efficacy outcome is the the difference between the active and sham treatment groups in morphine equivalence dosage.

DETAILED DESCRIPTION:
This is a single site, randomized, sham-controlled, double-blind study assessing the feasibility, safety, tolerability, and efficacy of non-invasive VNS (nVNS) in the treatment of headache in subarachnoid hemorrhage (SAH). The hypothesis is that two-two minute noninvasive stimulations of the cervical branch of the Vagus nerve, every 5 hours, is efficacious in safely reducing headache intensity and frequency in patients with headache due to SAH, during the patient's intensive care unit (ICU) stay. After screening and obtaining informed consent, eligible patients diagnosed with SAH on head scans, admitted to the Neurosurgical Intensive Care Unit (NSCU) at Northshore University Hospital will be randomized to either the treatment (stimulation of the cervical branch of the Vagus nerve) or sham (inactive stimulation) group. Pain intensity will be evaluated every 4 hours. Non-invasive stimulation will be performed every 5 hours. Device related adverse events, mean headache intensity, and mean and peak morphine equivalence dosage during the study period will be compared between the VNS group and the sham group.

The primary objective of this study is to examine the safety and effectiveness of nVNS as a treatment for headache in subarachnoid hemorrhage (SAH).

The primary safety endpoint for this study is the incidence of device related serious adverse events.

The primary outcome measurements for effectiveness is the difference between the active and sham treatment groups in morphine equivalence dosage

Secondary endpoints include descriptive comparisons between the active and sham treatment groups in:

* The difference between the active and sham treatment groups in the mean daily headache intensity
* The difference between total overall morphine equivalence dosage between the active and sham group per subject during study
* Opiate related adverse events (such as urinary retention, constipation, sedation, respiratory depression, nausea, vomiting and pruritis)
* The difference in CSF and blood inflammatory markers before and after VNS
* Difference in vessel diameter during angiogram for cerebral vasospasm before and after VNS

Study period is 14 days starting 24-72 hours post successful treatment of the aneurysm and extubation.

ELIGIBILITY:
Inclusion Criteria:

* Established signed and dated informed consent form
* CT of the head revealing blood in the subarachnoid space
* Subject is male or female, 18 to 80 years of age
* Subject alert to be able to verbalize pain level. If alertness improves after placement of an external ventricular drain, or once extubated, and the patient becomes alert , the patient will be enrolled
* Subject reports pain of > =7 on 10 Point Pain numeric rating scale
* Female of reproductive age must have a negative pregnancy test (Urine or blood test)

Exclusion Criteria:

* Use of any concomitant electrostimulation devices (Pacemaker, defibrillator, deep brain stimulation.)
* Unsecured aneurysm defined as aneurysm that has not been surgically or endovascularly treated.
* Previous carotid surgeries or known history of carotid artery disease
* Screws, metals or device in the neck
* History of secondary or tertiary heart blocks, ventricular tachycardia, Supra-Ventricular Tachycardia (including atrial fibrillation)
* Alcoholics (CAGE scale of 2 or greater). If patients are on Clinical Institute Withdrawal Assessment for Alcohol (CIWA) protocol for alcohol withdrawal, the patient will be excluded from the study.
* Drug addicts or chronic opioid users confirmed by history or with urine toxicology showing opiates or cocaine
* small traumatic SAH

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northshore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magalhaes JE, Azevedo-Filho HR, Rocha-Filho PA. The risk of headache attributed to surgical treatment of intracranial aneurysms: a cohort study. Headache. 2013 Nov-Dec;53(10):1613-23. doi: 10.1111/head.12165. Epub 2013 Jun 28. PMID 23808965
- [Background] Rumalla K, Smith KA, Arnold PM, Mittal MK. Subarachnoid Hemorrhage and Readmissions: National Rates, Causes, Risk Factors, and Outcomes in 16,001 Hospitalized Patients. World Neurosurg. 2018 Feb;110:e100-e111. doi: 10.1016/j.wneu.2017.10.089. Epub 2017 Oct 26. PMID 29107164
- [Background] Glisic EK, Gardiner L, Josti L, Dermanelian E, Ridel S, Dziodzio J, McCrum B, Enos B, Lerwick P, Fraser GL, Muscat P, Riker RR, Ecker R, Florman J, Seder DB. Inadequacy of Headache Management After Subarachnoid Hemorrhage. Am J Crit Care. 2016 Mar;25(2):136-43. doi: 10.4037/ajcc2016486. PMID 26932915
- [Background] Morad AH, Tamargo RJ, Gottschalk A. The Longitudinal Course of Pain and Analgesic Therapy Following Aneurysmal Subarachnoid Hemorrhage: A Cohort Study. Headache. 2016 Nov;56(10):1617-1625. doi: 10.1111/head.12908. Epub 2016 Oct 5. PMID 27704534
- [Background] Dorhout Mees SM, Bertens D, van der Worp HB, Rinkel GJ, van den Bergh WM. Magnesium and headache after aneurysmal subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2010 May;81(5):490-3. doi: 10.1136/jnnp.2009.181404. Epub 2009 Oct 13. PMID 19828484
- [Background] Oshinsky ML, Murphy AL, Hekierski H Jr, Cooper M, Simon BJ. Noninvasive vagus nerve stimulation as treatment for trigeminal allodynia. Pain. 2014 May;155(5):1037-1042. doi: 10.1016/j.pain.2014.02.009. Epub 2014 Feb 14. PMID 24530613
- [Background] Akerman S, Simon B, Romero-Reyes M. Vagus nerve stimulation suppresses acute noxious activation of trigeminocervical neurons in animal models of primary headache. Neurobiol Dis. 2017 Jun;102:96-104. doi: 10.1016/j.nbd.2017.03.004. Epub 2017 Mar 9. PMID 28286178
- [Background] Frangos E, Komisaruk BR. Access to Vagal Projections via Cutaneous Electrical Stimulation of the Neck: fMRI Evidence in Healthy Humans. Brain Stimul. 2017 Jan-Feb;10(1):19-27. doi: 10.1016/j.brs.2016.10.008. Epub 2016 Oct 20. PMID 28104084
- [Background] Bosche B, Graf R, Ernestus RI, Dohmen C, Reithmeier T, Brinker G, Strong AJ, Dreier JP, Woitzik J; Members of the Cooperative Study of Brain Injury Depolarizations (COSBID). Recurrent spreading depolarizations after subarachnoid hemorrhage decreases oxygen availability in human cerebral cortex. Ann Neurol. 2010 May;67(5):607-17. doi: 10.1002/ana.21943. PMID 20437558
- [Background] Chen SP, Ay I, Lopes de Morais A, Qin T, Zheng Y, Sadeghian H, Oka F, Simon B, Eikermann-Haerter K, Ayata C. Vagus nerve stimulation inhibits cortical spreading depression. Pain. 2016 Apr;157(4):797-805. doi: 10.1097/j.pain.0000000000000437. PMID 26645547
- [Background] Pavlov VA, Wang H, Czura CJ, Friedman SG, Tracey KJ. The cholinergic anti-inflammatory pathway: a missing link in neuroimmunomodulation. Mol Med. 2003 May-Aug;9(5-8):125-34. PMID 14571320
- [Background] Suzuki T, Takizawa T, Kamio Y, Qin T, Hashimoto T, Fujii Y, Murayama Y, Patel AB, Ayata C. Noninvasive Vagus Nerve Stimulation Prevents Ruptures and Improves Outcomes in a Model of Intracranial Aneurysm in Mice. Stroke. 2019 May;50(5):1216-1223. doi: 10.1161/STROKEAHA.118.023928. PMID 30943885
- [Background] George MS, Ward HE Jr, Ninan PT, Pollack M, Nahas Z, Anderson B, Kose S, Howland RH, Goodman WK, Ballenger JC. A pilot study of vagus nerve stimulation (VNS) for treatment-resistant anxiety disorders. Brain Stimul. 2008 Apr;1(2):112-21. doi: 10.1016/j.brs.2008.02.001. Epub 2008 Mar 28. PMID 20633378
- [Background] Breit S, Kupferberg A, Rogler G, Hasler G. Vagus Nerve as Modulator of the Brain-Gut Axis in Psychiatric and Inflammatory Disorders. Front Psychiatry. 2018 Mar 13;9:44. doi: 10.3389/fpsyt.2018.00044. eCollection 2018. PMID 29593576
- [Background] Lendvai IS, Maier A, Scheele D, Hurlemann R, Kinfe TM. Spotlight on cervical vagus nerve stimulation for the treatment of primary headache disorders: a review. J Pain Res. 2018 Aug 27;11:1613-1625. doi: 10.2147/JPR.S129202. eCollection 2018. PMID 30214271

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Arm | Treatment Group
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: active VNS group
- Sham: sham group ( no real stimulation)
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13) | 51 (11) | 52.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 7 | 6 | 13
mfs [Number; unit: participants] — Population: MODIFIED RANKIN SCALE IS A RANK FROM 1-4
  1. MEANS THIN BLOOD WITH NO IVH
  2. MEANS THIN BLOOD WITH IVH
  3. MEANS THICK CLOOD WITH IVH
  4. MEANS THICK BLOOD WITH IVH THE HIGHEST THE mFS the more blood there
  participants
    MFS1 | 4 | 2 | 6
    MFS2 | 1 | 2 | 3
    MFS3 | 8 | 9 | 17
    MFS4 | 6 | 8 | 14
HHS [Number; unit: participants] — Hunt Hess Scale Is a prognostic scale, how the patient presented on admission, the higher the scare the poorer the prognosis HHS1. no/mild headache HHS2, mod/seve headache, CN palsy HHS3, drowsy, min neuron deficit HHS4 Stupor,mod/sev hemiparesis HHS5- Deep coma, decerebrate Population: 40 overall , 21 in sham and 19 in active
  participants
    hhs1 | 5 | 7 | 12
    hhs2 | 10 | 11 | 21
    hhs3 | 2 | 2 | 4
    hhs4 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between the Active and Sham Treatment Groups in Morphine Equivalence Dosage PER DAY
Description: Daily morphine equivalence dosage will be calculated and compared between the active and Sham group
Time Frame: up to 14 days of admission
Population: 4O PARTICIPANTS , 19 IN ACTIVE GROUP AND 21 IN SHAM GROUP
Measure: Least Squares Mean (Standard Deviation); unit: mg
Groups:
- Active Device: received stimulation
- Sham: did not receive real stimulation
Arm/Group | Active Device | Sham
Number analyzed (Participants) | 19 | 21
mg | 0.058 (0.31) | 0.24 (0.29)

2. Primary Outcome: Overall Difference in MED at 7 Days
Description: difference in mean morphine equivalent dosage at 7 days between active and sham group
Time Frame: baseline and 7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Device | Sham
Number analyzed (Participants) | 19 | 21
mg | 21.99 (21.41) | 24.29 (14.5)

3. Secondary Outcome: The Difference Between the Active and Sham Treatment Groups in the Mean Daily Headache Intensity Pre and Post Stimulation
Description: Headache intensity is measured every 4 hours per standard of care. The pain intensity is reported using a 0 to 10 numeric rating scale, o being no pain, and 10 being severe pain. least mean square difference between the 2 groups between the pre and post stimulation pain score
Time Frame: up to 14 days of admission
Population: 40, 19 ACtIVE AND 21 SHAM
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- ACTIVE DEVICE: ACTIVE
- Sham: did not receive stimulation
Arm/Group | ACTIVE DEVICE | Sham
Number analyzed (Participants) | 19 | 21
units on a scale | -0.59 (0.11) | -0.13 (0.11)

4. Secondary Outcome: The Difference in Device Related Heart Rate Change Before and After Stimulation
Description: difference in change in Heart rate between the 2 groups from before to after stimulation
Time Frame: up to 14 days of admission
Population: between sham and active hear rate
Measure: Least Squares Mean (Standard Error); unit: beats per min
Groups:
- ACTIVE GROUP: received stimulation
- Sham: no stimulation
Arm/Group | ACTIVE GROUP | Sham
Number analyzed (Participants) | 19 | 21
beats per min | -1.73 (1.13) | -0.76 (1.18)

5. Secondary Outcome: Change in SBP Between Active and Sham Group
Description: difference between pre and post stimulation SBP between the 2 groups
Time Frame: before and after stimulation, up to 14 days
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury
Arm/Group | Active | Sham
Number analyzed (Participants) | 19 | 21
millimeters of mercury | -2.20 (0.88) | -1.64 (1.05)

ADVERSE EVENTS:
Time Frame: through study completion, up to 14 days
Description: Difference in Heart rate, SBP, DBP between the active and sham between before and after stimulation rate of VNS related side effects: skin irritation, hoarseness, dyspepsia, shortness of breath , arrhythmia between the two groups
Arm/Group | Sham Arm | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 5/21 | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Arm (N=21) | Treatment Group (N=19)
site discomfort (General disorders) | 0 (0) | 6 (6) — discomfort during stimulation
tingling sensation (General disorders) | 5 (5) | 9 (9) — tingling during stimulation
pain at stimulation (General disorders) | 2 (2) | 6 (6) — pain during stimulation
muscle twitching (General disorders) | 2 (2) | 8 (8) — twitching during stimulation
transient facial droop (General disorders) | 0 (0) | 6 (6) — during stimulation
dizziness (Nervous system disorders) | 0 (0) | 2 (2) — dizziness during stimulation
hoarseness (Ear and labyrinth disorders) | 2 (2) | 5 (5) — transient hoarseness during stimulation
dysgusia (General disorders) | 0 (0) | 0 (0) — dysgusia during stimulation
dyspnea (General disorders) | 0 (0) | 1 (1) — transient dyspnea during stimulation
nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) — nausea during stimulation
coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — coughing during stimulation
hoarseness (Ear and labyrinth disorders) | 0 (0) | 0 (0) — hoarseness during stimulation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04126408/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04126408/SAP_002.pdf